CLINICAL TRIAL: NCT05215808
Title: A First-in-Human, Randomized, Placebo-Controlled, Phase 1 Single and Multiple Ascending Dose Study to Assess the Safety and Pharmacokinetics of RBN-3143 in Healthy Subjects and as Open-Label in Patients With Atopic Dermatitis Subjects
Brief Title: SAD/MAD Safety and PK Study of RBN-3143 in Healthy and Atopic Dermatitis Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ribon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: RBN-3143-21-001
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Atopic Dermatitis
Keywords: Normal Healthy Volunteers; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: single dose ascending cohorts followed by multiple dose ascending cohorts
Who Masked: Participant, Care Provider, Investigator
Masking Description: 3:1 Randomization ratio of RBN-3143 to Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RBN-3143 (Experimental): RBN-3143 in single ascending dose followed by multiple ascending dose cohorts, randomized 3:1 ratio
  Interventions: Drug: RBN-3143
- Placebo (Active Comparator): Placebo randomized in 1:3 ratio with ascending RBN-3143 single and multiple dosing
  Interventions: Drug: RBN-3143
- Pantoprazole (Other): Open Label PPI cohort to evaluate concurrent administration of pantoprazole on RBN-3143 pharmacokinetics
  Interventions: Drug: RBN-3143
- Midazolam (Other): Open Label DDI Cohort (12 subjects) to evaluate the effect of RBN-3143 on the exposure of midazolam, a sensitive CYP3A4 substrate
  Interventions: Drug: RBN-3143

INTERVENTIONS:
Drug: RBN-3143 — Oral Administration of tablets

SUMMARY:
RBN-3143 Background: PARP proteins are members of a family of seventeen ADP-ribosyltransferase (ART) enzymes that regulate cellular processes including gene expression, protein degradation, and multiple cellular stress responses. RBN-3143 is a PARP-14 inhibitor. PARP14 is over-expressed in tissues with inflammatory diseases. RBN-3143 is a novel, orally administered PARP14 inhibitor that was developed to be evaluated as therapy for a range of inflammatory diseases, with an initial focus on Atopic Dermatitis.

Study Overview: The study consists of 2 parts. Part A: This part of the study is being conducted in a clinical research unit (CRU) and is enrolling healthy adult subjects to determine the safety of RBN-3143; its absorption, metabolism, and excretion (what the body does to this drug); and will assess its potential pharmacodynamic properties (what the drug does to the body).

There are 3 subsections to this part of the study. The first segment was conducted in a double-blind manner (neither the investigator nor subject knew if placebo or RBN-3143 was given) to assess dosing regimens of RBN-3143 when taken in a fasted state (before food). The last two segments are currently recruiting and are Open Label (all subjects will receive RBN-3143) and will assess RBN-3143 when taken with food, with pantoprazole, a medication that decreases the amount of acid in the stomach, and with midazolam.

Part B: In early 2023 the second part of the study will be conducted in patients with moderate to severe atopic dermatitis to measure the pharmacodynamic activity of RBN-3143 and evaluate preliminary efficacy of 28 days administration of the study drug. All patients will receive the same dose of RBN-3143.

DETAILED DESCRIPTION:
The study consists of 2 parts.

Part A: This part of the study is being conducted in a clinical research unit (CRU) and will enroll healthy adult subjects to determine the safety of RBN-3143; its absorption, metabolism, and excretion (what the body does to this drug); and will assess its potential pharmacodynamic properties (what the drug does to the body).

There are 3 subsections to this part of the study. The first subsection has completed enrollment and the 2 open-label subsections are now actively enrolling.

1. Double-Blind Cohorts- Fasting: In the first segment of the study, subjects were randomized in a double-blind manner using a 3:1 ratio (RBN-3143: placebo) to receive either RBN-3143 or placebo. Subjects were enrolled in groups of ascending doses.
2. Open Label Cohorts:

   1. Food Effect/Proton Pump Inhibitor (FE/PPI) Open Label Cohort:

      Twelve (12) additional subjects are being enrolled and will receive RBN-3143 with food (fed), fasted, or with pantoprazole, PPI, a drug to determine if the amount of acid in the stomach, as well as the presence or absence of food changes how RBN-3143 is absorbed. Subjects will be required to stay in the CRU for up to 16 days. Two sequences will be studied, either fasted then fed or fed then fasted with both sequences followed by administration of a proton pump inhibitor.
   2. Drug-Drug Interaction (DDI) Open Label Cohort: A further 12 subjects are being enrolled into a DDI cohort, to evaluate the effect of RBN-3143 on the exposure of midazolam, a sensitive CYP3A4 substrate. Subjects will be required to stay in the CRU 19 days. Subjects will also return for a final visit approximately 1 week later. This cohort will have 2 Treatment Periods as follows:

      * Treatment Period 1: On Day 1, subjects will be administered a single oral dose of 2 mg midazolam in the fasted state.
      * Treatment Period 2: Subjects will be administered RBN-3143 in the fasted state from Day 3 through Day 17 (14- day treatment period). On Day 16, subjects will also receive a single oral dose of 2 mg midazolam in the fasted state.

Part B: In early 2023 the second part of the study will be initiated in approximately 12 patients with moderate to severe atopic dermatitis. All patients will receive the same doses of RBN-3143 for 28 days.

On Day 1 and Day 28 patients will fast overnight until after the morning dose administration then fast for 4 hours post-dose. On all other days fasted state will be 2 hours prior to dosing and 2 hours after dosing. Patients will be required to present at the CRU on Day -1 for required study assessments after which they may return home. Patients will return to the CRU on Day 1 for the day 1 dose and the completion of required study assessments. Patients will then return home with sufficient study drug to complete dosing on Days 2 to Day 27 (inclusive). Patients will be required to attend the CRU for completion of required assessments on Day 7, Day 14, Day 21, and Day 28, and will return any remaining study drug on the Day 28 visit. Patients will return for an EOS/Follow-up visit at 4 weeks after the last dose of study drug.

Collection of data will cease at the time of database lock for final safety and PK analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects between 18 and 65 years of age (inclusive at the time of informed consent)
2. Body mass index (BMI) between ≥18 and ≤30 kg/m2 (inclusive) at Screening
3. Good general health, with no significant medical history, have no clinically significant abnormalities on physical examination at Screening and/or before administration of the initial dose of study drug
4. Clinical laboratory values within normal range as specified by the testing laboratory, unless deemed not clinically significant by the Investigator
5. Willingness and ability to speak, read, and understand English, and provide written informed consent
6. Must be a non-smoker or former smoker. Subjects must have negative cotinine results in drug tests at Screening and Baseline
7. Females must be:

   Non-pregnant Non-lactating Must use a non-hormonal, acceptable, highly effective double contraception from Screening until study completion, including the Follow-up Period

   Acceptable non-hormonal double contraception is defined as a condom AND one other form of the following:
   * An IUD (non-hormonal)
   * Documented evidence of surgical sterilization at least 6 months prior to Screening (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, or bilateral oophorectomy for women or vasectomy for men [with appropriate post-vasectomy documentation of the absence of sperm in semen] provided the male partner is a sole partner)

   Women of child-baring potential (WOCBP) must have:

   A negative pregnancy test at Screening and Day -1 and be willing to have additional pregnancy tests as required throughout the study

   Post-menopausal Women:

   Women not of childbearing potential must be:

   Postmenopausal for ≥12 months Postmenopausal status will be confirmed through testing of FSH levels ≥ 40 IU/L at Screening for amenorrhoeic female subjects

   Abstinence:

   Females who are abstinent from heterosexual intercourse will also be eligible. Complete abstinence by the subject for the duration of the study and for 1 month after the last study treatment is acceptable.

   Note: Periodic abstinence (eg, calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not considered highly effective methods of birth control.

   Female subjects who are in same-sex relationships are not required to use contraception.

   Males:

   If engaged in sexual relations with a WOCBP:

   The subject or his partner must be surgically sterile (eg, >30 days since vasectomy with no viable sperm, tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy)

   Must use an acceptable, highly effective contraceptive method from Screening until study completion, including the Follow-up Period. Acceptable methods of contraception include the use of condoms and the use of an effective contraceptive for the female partner that includes:
   * OCPs
   * Long acting implantable hormones
   * Injectable hormones
   * Vaginal ring
   * Use of an IUD

   Subjects with same-sex partners (abstinence from penile-vaginal intercourse) are eligible
8. For at least 90 days after the last dose of study drug, male subjects must not donate sperm and female subjects must not donate ovum
9. Willingness to comply with the drawing of all blood samples for the PK/PD analysis.
10. Willing and able to attend the necessary visits to the CRU and comply with all testing, fasting, and requirements defined in the protocol.
11. Willing and able to remain at the study site unite for the duration of the confinement period and return for outpatient visit/s defined in the protocol.

    FOR PART B (Moderate/Severe AD COHORT ONLY)

    In addition to the inclusion criteria stated above, patients must meet the following criteria for inclusion in Part B:
12. Chronic atopic dermatitis (AD) diagnosed by the Eichenfield revised criteria of Hanifin and Rajka, that has been present for at least 6 months before the Screening visit
13. EASI score ≥ 8 at the Screening and Baseline visits
14. IGA score ≥ 3 at the Screening and Baseline visits
15. Equal to or greater than 10% body surface area of AD involvement in areas affected beyond palms and soles at the Screening and Baseline visits, as per SCORAD
16. A documented history by the Investigator or delegate of inadequate response to treatment with topical medications within the past 6 months defined as failure to achieve or maintain remission or mild disease activity state (IGA score ≤ 2) despite daily treatment with topical corticosteroids of medium or higher potency (with or without topical calcineurin inhibitors) applied for at least 4 weeks or for the maximum recommended by the product manufacturer, whichever is shorter.
17. The patient must be applying stable doses of an additive-free, basic bland emollient twice-daily for at least 7 days before the Baseline visit
18. The patient must be willing to comply with skin biopsy/specimen collections

Exclusion Criteria:

1. Any medical condition that is considered by the Investigator or delegate that may interfere with study assessments, may adversely affect the subject's participation in the study, may make the subject's participation in the study unreliable, or be of such severity as to present an increased risk to the subject because of participation in the study.
2. Prior or ongoing medical conditions, physical findings, laboratory abnormality or a history of neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, or metabolic disease that is considered as significant by the Investigator or delegate, and in the Investigator's opinion, could adversely affect the safety of the subject
3. Abnormal ECG findings at Screening that are considered by the Investigator to be clinically significant:

   1. Significant history of cardiovascular disease
   2. ECG results showing QTcF >450 msec or the presence of clinically significant abnormalities as determined by the investigator (Screening or Day -1)
   3. Elevation of blood pressure (BP), i.e., supine systolic BP >140 mmHg and/or diastolic BP >90 mmHg, or heart rate >100 beats per minute at rest
4. Use of any prescription medication within 14 days of dosing or over-the-counter (OTC) medication (including vitamins) within 48 hours of dosing or intends to use any prescription medication or OTC medication during the study that may interfere with the evaluation of study medication. Co-administration of medications known to have high risk of prolonging the QT interval are also prohibited. The use of other concomitant medications that present a low risk of QT prolongation may be considered, with the approval of the Medical Monitor. Simple analgesia (paracetamol, nonsteroidal anti-inflammatory drug [NSAID]) may be permitted at the discretion of the Investigator or delegate. Use of a low dose corticosteroid and β2 agonist inhalers to treat concomitant Asthma are allowed.
5. Ingestion of herbal medicines within 3 weeks before Screening, and grapefruit, grapefruit juice, star fruit or orange marmalade (made with Seville oranges) within 2 weeks prior to dosing, or intends to use any of these products during the study
6. Relevant dietary restrictions or unwilling to consume standard meals provided.
7. Ingestion of caffeine- or xanthine-containing products (e.g., coffee, tea, cola drinks, and chocolate) on days scheduled for full PK sample collection from 10 hours prior to the start of dosing through 12 hours post-dose. Must refrain from the consumption of alcohol for 2 days prior to Day 1 through the end of the study
8. A history of substance abuse or dependency or history of recreational intravenous (IV) drug use over the last 1 year (by self-declaration); or a positive ethanol breath test, urine cotinine, or urine drug screen at Screening and at Day -1
9. A positive test for hepatitis C antibody (HCV), hepatitis B surface antigen (HBsAg), human immunodeficiency virus (HIV) antibody, or COVID-19 (if conducted, at the Investigator's discretion) at Screening
10. Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the Follow-up Period
11. Use of any investigational product (IP) or investigational medical device within 30 days prior to Screening, or 5 half-lives of the product (whichever is the longest) or participation in more than 4 investigational drug studies within 1 year prior to Screening
12. Donated or lost a significant volume of blood (>450 mL) within 4 weeks prior to the first study drug administration
13. Unwilling to reside in the study unit for the duration of the study or to cooperate fully with the Investigator, delegate or site personnel.
14. Alkaline phosphatase (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), and/or total bilirubin >1.5 × upper limit of normal at Screening. Repeat testing at Screening is acceptable for out-of-range values following approval by the Investigator or delegate
15. Estimated Glomerular Filtration Rate (eGFR) < 90 mL/min/1.73m2
16. Presence of any underlying physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the subject will comply with the protocol or complete the study per protocol
17. Plasma donation within 7 days prior to the first study drug administration
18. Fever (temperature >38°C) or symptomatic viral or bacterial infection within 2 weeks prior to Screening
19. History of severe allergic or anaphylactic reactions to medicines or vaccines
20. History of malignancy, except for non-melanoma skin cancer, excised more than 2 years ago and cervical intraepithelial neoplasia that has been successfully cured more than 5 years prior to Screening
21. History or presence of a condition associated with significant immunosuppression
22. History of life-threatening infection (e.g., meningitis)
23. Infections requiring parenteral antibiotics within the 6 months prior to Screening
24. For the Food effect cohort only: a diet that in the opinion of the Investigator is incompatible with the on-study diet (e.g., lactose intolerance diet)
25. Unwilling to refrain from strenuous exercise within 48 hours prior to visits and during confinement at the CRU

    FOR PART B (AD COHORT ONLY)

    In addition to the exclusion criteria stated above, patients must not enter Part B if any of the following exclusion criteria apply:
26. Use of any IP or investigational medical device within 8 weeks prior to Screening, or participation in more than 2 investigational drug studies within 1 year prior to Screening
27. Estimated Glomerular Filtration Rate (eGFR) < 60 mL/min/1.73 m2 at Screening
28. Vaccination with a live (attenuated) vaccine within 8 weeks before the Baseline visit
29. Treatment with allergen immunotherapy within 6 months before Screening
30. Treatment with leukotriene inhibitors within 4 weeks before the Baseline visit
31. Treatment with systemic corticosteroids within 4 weeks before the Baseline visit
32. Treatment with topical corticosteroids, tacrolimus, and/or pimecrolimus within 1 week before the Baseline visit
33. Systemic treatment for AD with an immunosuppressive or immunomodulating substance, eg, cyclosporine, mycophenolate-mofetil, IFN-γ, phototherapy (narrow band ultraviolet B [NBUVB], ultraviolet B [UVB], ultraviolet A1 [UVA1], psoralen + ultraviolet A [PUVA]), azathioprine, methotrexate, within 4 weeks before the Baseline visit and within 8 weeks for biologics
34. Use of any concomitant medication that is a moderate or strong inhibitor or inducer of CYP3A4 unless stopped 14 days prior to start of study treatment. Please refer to Section 28 (Appendix 1) for examples of such medications.
35. Use of any concomitant medication that is an inhibitor or inducer of P glycoprotein (P-gp) unless stopped 14 days prior to the start of study treatment. Please refer to Section 28 (Appendix 1) for examples of such medications.
36. Use of any concomitant medication that is a sensitive substrate of CYP3A4 and that, if underdosed, would constitute a significant risk to the subject. Individual cases may be discussed with the MM. Please refer to Section 28 (Appendix 1) for examples of such medications.
37. Use of a necessary concomitant medication where the exposure is dependent on drug transporters organic anion transporting polypeptide1B3 (OATP1B3) or multidrug and toxin extrusion protein 1 or 2-K (MATE1, MATE2-K) and that if overdosed would constitute a significant risk to the patient. Individual cases may be discussed with the MM
38. Subjects who have failed prior systemic treatment to selective inhibitor agents that regulate the interleukin signaling pathway (eg, dupilumab, JAK1 inhibitors except for veracitinib)
39. Treatment of AD with active medications (eg, Atopiclair®, MimyX®, Epicerum®, Cerave®, etc) within 1 week before the Baseline visit
40. Chronic or acute infection requiring treatment with oral or IV antibiotics, anti-virals, anti-parasitics, anti-protozoals, or anti-fungals within 4 weeks before the Baseline visit, or superficial skin infections within 1 week before the Baseline visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety determined by DLTs | 30 days
  Incidence rate of Dose limiting Toxicities (DLTs) of RBN 3143

SECONDARY OUTCOMES:
Cmax of RBN-3143 | Predose through 72 hours
  Assessment of maximum plasma concentration (Cmax) of RBN-3143
Tmax of RBN-3143 | Predose through 72 hours
  Time to maximum plasma concentration (Tmax)
AUC of RBN-3143 | Predose through 72 hours
  Assessment of area under the curve (AUC)
T1/2 of RBN-3143 | Predose through 72 hours
  Assessment of terminal half-life (T1/2)
CYP3A4 Assessment | Through Day 19
  Evaluate the effect of RBN-3143 on the exposure of midazolam
QTc | Predose through Day 7
  Assessment of corrected QT intervals via Fridericia's formula

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Polasek, MD, Principal Investigator — CMAX Clinical Research Pty Ltd
Locations (6):
- Australia (2):
  - Veracity Clinical Research, Woolloongabba, Queensland
  - CMAX Clinical Research Pty Ltd, Adelaide
- New Zealand (4):
  - Optimal Clinical Trials, Auckland
  - Waitemata Clinical Research, Auckland
  - New Zealand Clinical Research (NZCR), Christchurch
  - Southern Clinical Trials Tasman, Nelson

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caprara G, Prosperini E, Piccolo V, Sigismondo G, Melacarne A, Cuomo A, Boothby M, Rescigno M, Bonaldi T, Natoli G. PARP14 Controls the Nuclear Accumulation of a Subset of Type I IFN-Inducible Proteins. J Immunol. 2018 Apr 1;200(7):2439-2454. doi: 10.4049/jimmunol.1701117. Epub 2018 Mar 2. PMID 29500242
- [Background] Cho SH, Raybuck A, Wei M, Erickson J, Nam KT, Cox RG, Trochtenberg A, Thomas JW, Williams J, Boothby M. B cell-intrinsic and -extrinsic regulation of antibody responses by PARP14, an intracellular (ADP-ribosyl)transferase. J Immunol. 2013 Sep 15;191(6):3169-78. doi: 10.4049/jimmunol.1301106. Epub 2013 Aug 16. PMID 23956424
- [Background] Cohen MS, Chang P. Insights into the biogenesis, function, and regulation of ADP-ribosylation. Nat Chem Biol. 2018 Feb 14;14(3):236-243. doi: 10.1038/nchembio.2568. PMID 29443986
- [Background] Goenka S, Boothby M. Selective potentiation of Stat-dependent gene expression by collaborator of Stat6 (CoaSt6), a transcriptional cofactor. Proc Natl Acad Sci U S A. 2006 Mar 14;103(11):4210-5. doi: 10.1073/pnas.0506981103. Epub 2006 Mar 6. PMID 16537510
- [Background] He H, Bissonnette R, Wu J, Diaz A, Saint-Cyr Proulx E, Maari C, Jack C, Louis M, Estrada Y, Krueger JG, Zhang N, Pavel AB, Guttman-Yassky E. Tape strips detect distinct immune and barrier profiles in atopic dermatitis and psoriasis. J Allergy Clin Immunol. 2021 Jan;147(1):199-212. doi: 10.1016/j.jaci.2020.05.048. Epub 2020 Jul 21. PMID 32709423
- [Background] Iwata H, Goettsch C, Sharma A, Ricchiuto P, Goh WW, Halu A, Yamada I, Yoshida H, Hara T, Wei M, Inoue N, Fukuda D, Mojcher A, Mattson PC, Barabasi AL, Boothby M, Aikawa E, Singh SA, Aikawa M. PARP9 and PARP14 cross-regulate macrophage activation via STAT1 ADP-ribosylation. Nat Commun. 2016 Oct 31;7:12849. doi: 10.1038/ncomms12849. PMID 27796300
- [Background] Mehrotra P, Hollenbeck A, Riley JP, Li F, Patel RJ, Akhtar N, Goenka S. Poly (ADP-ribose) polymerase 14 and its enzyme activity regulates T(H)2 differentiation and allergic airway disease. J Allergy Clin Immunol. 2013 Feb;131(2):521-31.e1-12. doi: 10.1016/j.jaci.2012.06.015. Epub 2012 Jul 25. PMID 22841009
- [Background] Mehrotra P, Krishnamurthy P, Sun J, Goenka S, Kaplan MH. Poly-ADP-ribosyl polymerase-14 promotes T helper 17 and follicular T helper development. Immunology. 2015 Dec;146(4):537-46. doi: 10.1111/imm.12515. Epub 2015 Sep 28. PMID 26222149
- [Background] Vyas S, Chesarone-Cataldo M, Todorova T, Huang YH, Chang P. A systematic analysis of the PARP protein family identifies new functions critical for cell physiology. Nat Commun. 2013;4:2240. doi: 10.1038/ncomms3240. PMID 23917125